项目来源与编号:

# 嵌合抗原受体 T 细胞免疫疗法(CAR-T)治疗 难治性膜性肾病的安全性和有效性研究

项目负责人: 何丽洁

承担科室: 肾脏内科

联系电话: 029-89661611

承办单位:空军军医大学第一附属医院

研究年限: 2025年08月01日-2028年07月31日

版本号: V3.0

版本日期: 2025年10月10日

# 目录

| 方 案 摘 要 | 1 |
|---------------------|----|
| 一、研究背景 | 4 |
| 二、研究目的 | 7 |
| 三、研究设计 | 7 |
| 四、病例选择 | 8 |
| 1.入选标准 | 8 |
| 2.排除标准 | 9 |
| 3.终止研究标准 | 11 |
| 五、研究方法与技术路线 | 12 |
| 1.干预措施 | 12 |
| 2.样本量确定 | 14 |
| 3.数据信息采集和随访 | 15 |
| (1) 收集的数据 | 15 |
| (2) 数据完整性 | 17 |
| 4.技术路线图 | 18 |
| 六、观察项目与检测时点 | 18 |
| 1.主要观察终点 | 18 |
| (1) 剂量限制性毒性 (DLT) | 19 |
| (2) 不良事件(AE) | 20 |
| 2.次要观察终点 | 21 |
| (1) rMN 缓解或复发情况 | 21 |
| (2) 肾功能、免疫特征及细胞动态变化 | 22 |

| | (3) 检测时点 | 22 |
|----|---------------------------------------|----|
| 七、 | 不良事件的观察与处理 | 24 |
| | (一) 淋巴细胞清除期 | 24 |
| | (二) CAR-T 细胞回输后 | 24 |
| | 1. 细胞因子释放综合征(CRS) | 25 |
| | 2. 免疫效应细胞相关神经毒性综合征(ICANS) | 26 |
| | 3. 免疫效应细胞相关噬血细胞性淋巴组织细胞增生症样综合征(IEC-HS) | 29 |
| | 4. CAR-T 相关出凝血性疾病(CARAC) | 32 |
| | 5. 免疫效应细胞相关血液毒性(ICAHT) | 33 |
| | 6. B 细胞缺乏症/低丙种球蛋白血症 | 34 |
| | 7. 感染 | 36 |
| | 8. 过敏反应 | 39 |
| | 9. CAR-T 细胞异常增殖 | 40 |
| 八、 | 研究的质量控制与质量保证 | 40 |
| 九、 | 统计学处理 | 40 |
| +, | 临床研究的伦理学 | 41 |
| +- | - 、研究进度 | 41 |
| += | 二、参考文献 | 42 |

# 方案摘要

| 项目名称 | 嵌合抗原受体 T 细胞免疫疗法(CAR-T)治疗难治性膜性肾病(rMN)的安全性和有效性研究 |
|---|---|
| 研究目的 | 初步评估 CD19 CAR-T 在 rMN 中的安全性和有效性,以期为优化疾病治疗和管理提供新思路 |
| 研究设计 | 本研究是一项由西京医院肾脏内科何丽洁副教授团队发起的为单中心小样本探索性试验。患者在接受 CAR-T 细胞治疗前接受环磷酰胺(必要时加用氟达拉滨)去淋巴化疗。在预防性应用抗组胺药物和对乙酰氨基酚后,给予 CD19 CAR-T (1×10%kg)细胞输注。在随后的2周,住院监测患者生命体征及不良反应,本研究计划随访时间2年。 |
| 病例总数 | 5 |
| 病例选择 | <ul> <li>入选标准:</li> <li>(1) 经肾活检确诊为原发性膜性肾病(PMN);</li> <li>(2) 中等风险或高风险的 rMN;</li> <li>(3) 年龄≥18 周岁的患者;</li> <li>(4) eGFR≥30 ml/min/1.73m²,且无严重心、肝、肺功能异常;</li> <li>(5) 签署书面知情同意书</li> </ul> |
| | <i>排除标准:</i> (1)继发性膜性肾病; |
| | (2)活动性细菌、真菌、病毒(非普通感冒/流感)感 |

| | 染需静脉抗生素治疗,或活动性肺结核,或乙肝病毒(HBV)、 |
|------|-----------------------------------|
| | 丙肝病毒 (HCV)、艾滋病毒 (HIV)、梅毒螺旋体 (TP)、 |
| | EB 病毒(EBV)或巨细胞病毒(CMV)血清学阳性; |
| | (3)严重合并症或基础疾病; |
| | (4) 恶性肿瘤史; |
| | (5)治疗史排除,符合下列任意一个条件: |
| | a. 既往接受过任何细胞治疗(如间充质干细胞 |
| | 等); |
| | b. 入组前 24 周接受大手术,或计划在入组后 24 |
| | 周内接受手术; |
| | c. 计划3年内进行肾移植; |
| | d. 药物滥用史。 |
| | (6)入组前3个月内参加过其他干预性临床试验; |
| | (7) 妊娠期、哺乳期女性; |
| | (8) 无法理解研究或提供知情同意(如严重痴呆、精神 |
| | 疾病); |
| | (9) 存在任何研究者认为可能增加风险、干扰评估或影 |
| | 响依从性的情况。 |
| | 主要接受的干预措施包括外周血单个核细胞采集、去淋巴化 |
| 干预措施 | 疗及自体 CAR-T 注射液回输 |
| | 主要终点:安全性评价,以单次 CART 输注后的剂量限制性 |
| 评定 | 毒性(DLT)和不良事件(AE)的类型和发生率为评价指标 |
| | 次要终点:有效性评价: ①rMN 缓解或复发情况。细胞输注 |

| | 后维持缓解或部分缓解的受试者比例、缓解的持续时间以及 |
|---|---|
| | 复发;②肾功能、免疫特征及细胞动态变化,包括蛋白尿、 |
| | eGFR、血清抗 PLA2R 抗体、感染指标、补体、免疫球蛋白、 |
| | 细胞因子水平变化、外周血免疫细胞亚群变化, CD19 在外 |
| | 周血B细胞亚群表面的表达水平等。 |
| 统计方法 | 所有统计分析都不考虑受试者依从性差、中途退出或失访等情况。由于本研究样本量较小,所有数据均以个体数值呈现。研究将采用描述性统计方法报告基线期和随访期的特定参数,统计分析和数据展示使用 SPSS 27.0 和 GraphPad Prism9.0 版本完成。 |
| 研究期限 | 2025年08月-2028年07月 |

#### 一、研究背景

原发性膜性肾病(Primary Membranous Nephropathy, PMN)是一种由自身反应性 B 淋巴细胞产生的致病性抗体介导的自身免疫性疾病。这些抗体经血液循环到达肾脏,与肾小球基底膜上的特异性抗原结合形成原位免疫复合物。这些复合物继而引发一系列病理效应,最终导致肾小球足细胞损伤及大量蛋白尿[1]。目前全球 PMN 发病率约为 8-10 人/百万人[2],我国报告的发病率为 23.4%[3],PMN 的具体病因仍然未知,而其余病例与药物使用或系统性红斑狼疮、乙型肝炎病毒或恶性肿瘤等潜在疾病有关。尽管约三分之一的患者可能通过保守治疗实现自发完全或部分缓解,但另外三分之一患者面临疾病进展风险增加,可能在 10 年内导致终末期肾病[4]。

近十余年来,PMN的发病机制与治疗策略研究取得了显著进展。目前已鉴定出十余种与其相关的靶抗原,其中约70%的病例由抗磷脂酶 A2 受体(PLA2R)抗体介导<sup>[5]</sup>。针对抗体产生这一核心病理环节,当前的主要治疗策略是靶向清除产生自身抗体的B细胞及其终末分化的浆细胞<sup>[6]</sup>。以利妥昔单抗(Rituximab, RTX)为代表的抗CD20单克隆抗体是目前临床治疗PMN应用较广泛的靶向药物。其作用机制为特异性结合B细胞表面的CD20蛋白,从而清除B细胞,虽然RTX等被认为对PMN患者安全有效,但其有效性仍有局限,因为约30%的患者没有反应,这种反应不足可能是由于PLA2R抗体滴度较高<sup>[7]</sup>。此外,部分患者在接受RTX治疗后会产生抗药物抗体,也可

能导致药物清除加速、疗效降低(耐药)或疾病复发<sup>[8]</sup>。此类难治性膜性肾病(Refractory Membranous Nephropathy,rMN)患者,即对RTX治疗无应答(表现为蛋白尿长期不缓解),进展至终末期肾脏病(End-Stage Renal Disease, ESRD)的风险显著增高<sup>[9,10]</sup>。这类患者表现为:确诊时抗PLA2R 抗体阳性,在接受足量、足疗程的一线免疫抑制治疗后,抗PLA2R 抗体滴度持续处于高水平或无明显变化;或抗PLA2R 抗体虽持续阴性,但一线免疫治疗持续6个月以上肾病综合征仍未缓解的患者。因此,有必要探索疗效更好的替代疗法。

嵌合自身抗体受体 T 细胞 (CAR-T) 疗法通过白细胞分离术分离外周血中的单核细胞,然后在体外进行基因工程改造以表达嵌合抗原受体。因此, CAR-T 细胞无需抗原处理和呈递即可识别靶细胞上的特异性抗原。一旦经过基因改造, CAR-T 细胞就会在体外经历广泛增殖,用淋巴细胞耗竭化疗后,这些细胞被重新注入患者体内。该疗法的优点是机体会形成长期记忆 CAR-T 细胞,无需重复给药即可对新产生的靶细胞提供持续的疗效[11]。

因 CAR-T 疗法的靶向作用,其在临床的应用逐渐广泛,在自身免疫性疾病,包括肾脏疾病中也显示出较好的应用前景。2021 年 8 月首次报道了一例严重 SLE 患者接受 CD19 CAR-T 细胞治疗并取得较好疗效的病例<sup>[12]</sup>。随后,2022 年 9 月,该团队报道了另外 5 例接受 CD19 CAR-T 细胞治疗的难治性 SLE 患者,所有患者病情改善,狼疮性肾炎均达到临床治愈,血清补体、双链 DNA 抗体恢复正常<sup>[13]</sup>。2024 年 2 月,该团队发表了关于 CD19 CAR-T 治疗自身免疫性疾病

的研究结果,该研究纳入自身免疫性疾病患者 15 例,包括 8 名 SLE 患者,4 名系统性硬化症和 3 名特发性肌炎患者,这些患者有活动性器官受累迹象,经历至少两种免疫治疗方案失败,且其疾病严重,有危及生命可能,接受 CAR-T治疗随访 15 个月后,所有 8 名 SLE 患者均实现了疾病缓解,4 名系统性硬化患者疾病活动指数下降,特发性肌炎患者疾病也得到控制[14]。

在治疗免疫性疾病方面,CAR-T疗法的不良反应与血液系统肿瘤一致,最主要的为细胞因子释放综合征(CRS),其他可能出现的副作用包括免疫效应细胞相关神经毒性综合征(ICANS)、免疫效应细胞相关噬血细胞性淋巴组织细胞增生症样综合征(IEC-HS)、CAR-T相关出凝血性疾病(CARAC)、免疫效应细胞相关血液毒性(ICAHT)、B细胞缺乏症或低丙种球蛋白血症及感染等[15]。现有研究显示,CAR-T细胞疗法的急性毒性反应发生率低与程度轻,短期安全性良好,尤其是在自身免疫病中耐受性优异,主要风险为轻度 CRS 和可管控的感染,无治疗相关死亡或严重并发症(如无弥散性血管内凝血、多器官衰竭、需呼吸机支持等事件)[13,14,16-18]。总之,前期的 CAR-T细胞疗法在自身免疫性疾病小样本临床研究成果表明 CAR-T细胞疗法提示其在自身免疫性疾病中广阔的应用前景。

针对 MN 抗原特异性治疗方案的潜在靶点包括自身抗体产生、抗体-抗原相互作用和免疫介导的足细胞损伤<sup>[19]</sup>。在 rMN 中,阻碍抗体的产生显然具有关键意义。CAR-T 细胞疗法是一种流行的策略,不仅可以消灭特定的致病性抗原及其表位(如 CD19<sup>+</sup>B 细胞),还可以

在体内产生具有记忆的 CAR-T 细胞,实现长期持续清除的潜力<sup>[20]</sup>。因此,我们的研究目的是通过前瞻性、小样本临床试验初步评估 CD19 CAR-T 疗法在 rMN 中的安全性及有效性,以期为 rMN 提供更好的治疗策略。

# 二、研究目的

当前,rMN 患者对于一线免疫或靶向治疗无应答,进展为终末期肾脏病的风险显著增高。因此,仍需进一步探索 rMN 的有效治疗手段。CAR-T 细胞在自身免疫性疾病临床研究中的成果提示其在 rMN 中可能具有较好的潜力与应用前景。因此,我们的研究目的是通过前瞻性、小样本临床试验初步探索 CAR-T 疗法在 rMN 中的安全性及有效性,以期为 rMN 提供更好的治疗策略。

# 三、研究设计

患者在自体 CAR-T 细胞治疗前 1-4 周期间进行外周血单个核细胞 采集,由陕西医赛尔生物科技有限公司(Shaanxi Yisaier Biotechnology Co., Ltd)完成分选纯化、T 细胞激活、CAR 基因转导、CAR-T 细胞体外扩增,经清洗、制剂、冻存、检测、放行环节后,再以冷链运输到层流病房进行静脉输注。所有患者在接受 CAR-T 细胞治疗前 3-7 天需进行去淋巴化疗重构免疫环境,首选方案为环磷酰胺(CTX)400mg/d,连续两天,第三天检测外周血淋巴细胞清除程度,若清除效果不佳,予以氟达拉滨(Flu)25 mg/m²/d,1~2 天。去淋巴化疗后>2 天,予以 CD19 CAR-T(1×106/kg)回输,细胞静脉输注前预防性应用抗组胺药物(如氯苯那敏或苯海拉明)和对乙酰氨

基酚。所有患者在层流病房至少住院观察 10 天,出现 3 级以上细胞因子释放综合征(CRS)等严重不良事件患者延长至 14 天。整个研究计划随访周期为 1 年,研究结束后的超长期随访将一直进行。

研究期间,每名受试者入组时间间隔不少于28天。

# 四、病例选择

# 1.入选标准

- 1) 经肾活检确诊为原发性膜性肾病(PMN);
- 2) 中等风险或高风险的 rMN;
  - a. 中等风险定义: eGFR ≥90 ml/min/1.73m², 24 小时尿蛋白>3.5g/d,接受肾素血管紧张素系统抑制剂(RASi)的6个月内尿蛋白下降不大于50%;
  - b. 高风险定义: eGFR<60ml/min/1.73m²和/或蛋白尿持续6个月以上>8g/d,或者 eGFR 正常,蛋白尿>3.5g/d,在接受 RASi的6个月尿蛋白下降不大于50%,并且至少满足下列任意一个条件:
    - ◆血清白蛋白<25g/L,
    - ◆PLA2Rab>50 RU/mI,
    - ◆尿α<sub>1</sub> 微球蛋白>40 μ g/min,
    - ◆尿 IgG>1 µ g/min,
    - ◆尿β2微球蛋白>250mg/d,
    - ◆筛选系数(IgG 清除率/白蛋白清除率)>0.20;
  - c. rMN 定义为: 在接受足量、足疗程(≥6个月)的标准

- 一线免疫抑制治疗(包括但不限于:糖皮质激素+环磷酰胺(CTX)方案,或钙调磷酸酶抑制剂[CNI],或利妥昔单抗(RTX))后,满足以下任一:
  - ◆抗 PLA2R 抗体持续高滴度阳性或无显著下降;
  - ◆抗 PLA2R 抗体阴性者,持续表现为肾病综合征 (24 小时尿蛋白>3.5g,血清白蛋白<30g/L);
  - ◆24 小时尿蛋白下降 <50%。
- 3) 年龄≥18周岁的患者;
- 4) 关键器官功能满足以下要求:
  - ◆肾功能: eGFR≥30 ml/min/1.73m<sup>2</sup>;
  - ◆肝功能: ALT 和 AST≤2.5×正常上限值 (ULN), 总胆红素≤1.5×ULN;
  - ◆心功能: 左心室射血分数 (LVEF)≥50%, NYHA 心功能分级I或 II 级的心力衰竭; 无需临床干预 的严重心律失常(如室性心动过速、心室[房]颤动、III°房室传导阻滞等)。近6个月内无急性 冠脉综合征、卒中、主动脉夹层等心脑血管事件。
  - ◆呼吸功能: 非吸氧状态下指脉氧饱和度 > 92%
- 5) 充分理解研究目的、风险与获益,自愿参与并签署书面知 情同意书(本人及法定监护人,如适用)。

# 2.排除标准

1) 继发性膜性肾病(如 SLE、肿瘤、药物、感染等所致);

- 2) 活动性细菌、真菌、病毒(非普通感冒/流感)感染需静脉 抗生素治疗,或活动性肺结核,或病毒血清学阳性,符合 下列任意一个条件:
  - ◆HBsAg (+) 和/或 HBcAb (+) 且 HBV DNA > 检测下限;
  - ◆HCV Ab (+) 且 HCV RNA (+);
  - **♦**HIV Ab (+);
  - ◆活动性 EBV/CMV: EBV IgM (+) 或 EBV-DNA > 正常值; CMV IgM (+) 或 CMV-DNA > 正常值;
  - ◆梅毒螺旋体(TP)抗体阳性(需评估活动性)。
- 3) 严重合并症/基础疾病。如未控制的高血压(如收缩压 > 160mmHg 或 舒张压 > 100mmHg 持续);或未控制的糖尿病(HbA1c > 8% 或 随机血糖 ≥ 11.1 mmol/L)或糖尿病肾病;或近 6 个月内有症状性深静脉血栓或肺栓塞史;或近 6 个月内有活动性消化性溃疡和/或消化道出血史;或先天性或获得性严重免疫缺陷(如 HIV、原发性免疫缺陷病);或严重中枢神经系统疾病(如灾难性抗磷脂综合征、癫痫未控);或非 PMN 所致的终末期器官衰竭;
- 4) 恶性肿瘤史。除己治愈的皮肤基底/鳞状细胞癌、宫颈原位癌、甲状腺癌外,5年内有恶性肿瘤史;
- 5) 治疗史排除,符合下列任意一个条件:
  - ◆既往接受过任何细胞治疗(如间充质干细胞、造

血干细胞移植等);

- ◆入组前 24 周接受大手术,或计划在入组后 24 周内接受手术;
- ◆计划3年内进行肾移植;
- ◆药物滥用史。
- 6) 入组前3个月内参加过其他干预性临床试验;
- 7) 妊娠期、哺乳期女性;
- 8) 无法理解研究或提供知情同意(如严重痴呆、精神疾病);
- 9) 存在任何研究者认为可能增加风险、干扰评估或影响依从性的情况。

# 3.终止研究标准

研究受试者的退出标准包括:

- 1) 安全性事件。发生与研究治疗(如淋巴细胞清除化疗、 CAR-T 输注)相关的严重不良事件(SAE) 或 不可耐受 毒性,研究者判断需永久停止治疗;
- 2) 受试者意愿。受试者或其法定监护人主动要求退出研究;
- 3) 受试者失访或死亡。
- 4) 出现非 PMN 相关的严重并发症(如新发恶性肿瘤、严重感染),需优先处理。
- 5) PMN 病情急剧恶化(如急性肾损伤需透析),研究者判断 不官继续试验。
- 6) 研究者判断继续研究不符合受试者最佳利益(如治疗无效

且风险增加),或重大方案违背影响主要终点评估。

7) 监管机构或伦理委员会要求终止研究。

退出后处理:详细记录退出原因、日期、末次治疗情况,提供标准治疗并持续随访安全性和疗效(除非受试者拒绝),已收集数据在符合伦理前提下用于统计分析。

# 五、研究方法与技术路线

1.干预措施

所有患者均在接受标准对症和支持疗法的基础上,接受 CD19 CAR-T 细胞治疗。

(1) 对症和支持治疗

所有患者均接受可达最大耐受性的保守治疗,主要有:

- ①血压控制与肾功能保护药物。包括但不限于:肾素血管紧张素醛固酮系统抑制剂(RAASi)、其他治疗高血压的一线药物(如利尿剂、β 受体阻滞剂、CCBs、α 受体阻滞剂或中枢神经系统活性药物等)、和钠-葡萄糖协同转运蛋白 2 抑制剂 SGLT-2i;
- ②血脂调控药物。包括但不限于:他汀类、贝特类、依折麦布及 PCSK9 抑制剂等;
  - ③降尿酸药物。包括但不限于: 非布司他、别嘌醇等;
  - ④钙磷代谢调节剂。包括但不限于钙剂、骨化三醇等;
  - ⑤抗贫血药。包括但不限于铁剂、叶酸等;
  - ⑥其他必要的非免疫抑制或调节类药物。
    - (2) CD19 CAR-T 细胞治疗

所有患者接受单次 1×10<sup>6</sup>/kg 自体 CD19 CAR-T 细胞治疗,主要流程有:

- ①外周血单个核细胞采集。利用血液成分分离机采集患者的血液,分离含有 T 细胞的血液。预计采集血量体积为 120ml,最少不低于 50 ml。采集过程,血液流速设定在 50~70 ml/min,必要时,采集人员将根据实际收集情况调整收集速度,采集时间预计在 2~4 小时。
- ②淋巴细胞清除化疗。研究将采用 CTX ± Flu 方案, 经全面评估 患者状态,确认患者能够耐受淋巴细胞清除化疗后,予以 CTX 400 mg/d,静脉注射,连续两天,总剂量 800mg,第三天检测外周血淋巴 细胞清除程度,若清除效果不佳则追加 Flu 25 mg/m²/d, 1~2 天。
- ③自体 CD19 CAR-T 细胞注射液回输。回输前 30~60 分钟使用对乙酰氨基酚衍生物和抗组胺药物(如氯苯那敏或苯海拉明)等。 CD19 CAR-T 细胞注射液采用静脉途径回输治疗,使用不带滤网的输血管,以防止有效细胞成分的丢失而降低疗效。回输程序为:生理盐水 100 ml 冲管→细胞回输→生理盐水 100 ml 冲管,前 15min 回输速度控制在 2~3 ml/min,以确保患者耐受性,无不良反应时可改为 5~10 ml/min。



图 1 研究主要干预措施与流程

表 1 研究流程计划表

| 阶段 | 时间 | 关键活动 | 评估重点 |
|----------|--------|------------------------------|--------------------|
| 患者筛选 | -6~-4w | 病史审查、实验室检测、影像学检查 | 符合难治性 MN 标准,器官功能达标 |
| 细胞制备 | -4~-1w | 患者评估、单采白细胞、CAR-T 改造与扩增、质检 | 细胞活性与安全性合格 |
| 清淋预处理 | -7~-3d | 环磷酰胺±氟达拉滨方案 | 淋巴细胞清除,预防感染 |
| CAR-T 回输 | Day 0 | 静脉输注 CAR-T 细胞 | 输注反应监测 |
| 住院监测 | d0-d14 | CRS/ICANS 管理、感染预防、早期<br>疗效评估 | 急性毒性控制,B 细胞耗竭 |
| 密集随访 | ≤3m | 每月临床评估、实验室检查 | 肾脏应答,免疫指标 |
| 中长期随访 | 3~12m | 定期全面评估、免疫重建监测 | 无药缓解状态,复发迹象 |
| 超长期随访 | >12m | 复发率、远期副作用追踪 | 长期安全性,生存质量 |

# 2.样本量确定

该研究为临床 I 期探索性试验, 初步预计纳入 5 例 rMN 患者。

终点评估

AE 评估

# 3.数据信息采集和随访

# (1) 收集的数据

所有的受试者在不同的研究阶段需完成知情同意书签署、病史信 息、查体、心电图/心脏超声、肾脏评估、常规检查、伴随用药记录、 终点结局评估等数据信息的采集(表2),这些数据信息包括但不限 干:

- ① 人口学资料。包括姓名、性别、出生年月、民族、文化程度、 职业、婚姻状况、现住址、联系方式。
- ② 伴随用药记录。主要包括降压、调脂、降糖、免疫调节、辅助 治疗、疫苗接种等相关药物的使用情况。
- ③ 生命体征。主要包括心率、血压、体温等。

CART 制 住院随访 密集随访 中长期随 研究结 研究结束后随访 计划 基线期 筛选期 备期 期 期 访 (超长期随访) 束随访 -6 to -4 to -2d to d0 to 时间 ≪3m 3 to 12m 12y >12m -4 w $-1\mathbf{w}$ d0d14 知情同意 Χ 纳排标准 Χ 人口学资料 Χ 既往史 Χ 用药史 Χ 伴随用药 Χ Χ Χ Χ Χ Χ Χ Χ 杏体 Χ Χ Χ Χ 体重、身高 Χ Χ Χ Χ Χ Χ 生命体征 Χ Χ Χ Χ Χ Χ Χ Χ 心电图/心脏超声 Χ Χ 肾脏超声 Χ Χ 实验室检查 Χ Χ Χ Χ Χ Χ

表 2. 研究活动和评估时间表

Χ

# (2) 研究流程与随访计划

- ① 筛选阶段。根据纳排标准筛选潜在的受试者,符合纳入标准的受试者由患者本人或其法定代理人签署知情同意书,收集人口学信息、既往史、用药史、伴随用药、体格检查、生命体征等数据;完成术前十二导联心电图、心脏超声、肾脏超声;完善血尿便常规、肝肾功能、血脂、血糖、电解质、凝血功能、抗 PLA2R 抗体、感染筛查(HBV、HCV、梅毒、HIV、EBV、CMV等)、尿微量白蛋白/肌酐(UACR)及尿蛋白定量。
- ② CART 制备阶段。记录伴随用药情况、体格检查、生命体征等数据;完善血尿便常规、肝肾功能、血脂、电解质、凝血功能、感染筛查(HBV、HCV、梅毒、HIV、EBV、CMV等)。
- ③ 基线阶段。记录伴随用药情况、体格检查、生命体征等数据; 完善血尿便常规、肝肾功能、血脂、血糖、电解质、凝血功能、C 反 应蛋白(CRP)、降钙素原(PCT)、抗 PLA2R 抗体、铁蛋白、补 体、免疫球蛋白、细胞因子、外周血淋巴细胞亚群、外周血 CD19 B 细胞、UACR 及 24 小时尿蛋白定量等实验室检查;完成心电图检查。
- ④ 住院随访期。记录伴随用药情况、体格检查、生命体征等数据;完善血尿便常规、肝肾功能、电解质、凝血功能、CRP、PCT、抗 PLA2R 抗体、铁蛋白、补体、免疫球蛋白、细胞因子、外周血淋巴细胞亚群、外周血 CD19 B 细胞表达、CAR 拷贝参数、UACR 及24 小时尿蛋白定量等实验室检查

- ⑤ 密集随访阶段。共计划完成 3 次随访,在接受回输治疗的第 28 天,完成出院后第一次随访 (随访 1)。计划完成血尿常规、肝肾功能、凝血功能、CRP、PCT、抗 PLA2R 抗体、铁蛋白、补体、免疫球蛋白、细胞因子、外周血淋巴细胞亚群、UACR 及 24 小时尿蛋白定量等实验室检查。随后的第二次和第三次随访 (随访 2 和 3)分别为治疗后的第 2 和第 3 月,计划完成血尿常规、肝肾功能、抗 PLA2R抗体、补体、免疫球蛋白、外周血淋巴细胞亚群、外周血 CD19 B 细胞表达、CAR 拷贝参数、UACR 及 24 小时尿蛋白定量等实验室检查。每次随访也应记录伴随用药情况、生命体征等数据。
- ⑥ 中长期随访阶段。治疗后第3个月至第12个月间,每3个月完成一次随访,共计3次随访计划,分别为随访4(治疗后第6个月)、随访5(治疗后第9个月)和随访6(治疗后第12个月),其中随访6也是研究结束随访。每次随访计划完成血尿常规、肝肾功能、抗PLA2R 抗体、补体、免疫球蛋白、CAR 拷贝参数、UACR 及24小时尿蛋白定量等实验室检查。随访4还需要完成外周血淋巴细胞亚群、外周血CD19B细胞表达检测。每次随访也应记录伴随用药情况、生命体征等数据。
- ⑦ 超长期随访阶段。该随访阶段为研究后随访,不严格设置随访计划,建议患者每3至6月定期自行前往本中心或就近于当地医疗机构完成必要的实验室和影像学检查。研究团队将持续通过电话、短信、微信等形式持续随访患者基本生命体征与病情变化等情况。

# (2) 数据完整性

# ① 常规临床访视数据采集

本研究采用纸质版病例报告表(CRF)表进行数据采集,使用 Epidata 数据库进行数据管理,采用双录入比较法进行数据录入和校 验,并进行相应的数据校验和清理。在研究期间,原则研究人员将每 月检查一次试验数据,以确保内部一致性。

# ② 向受试者发送提醒消息

将通过微信群、短信或电话提前向受试者发送自动提醒信息,从 而最大限度地减少因失访和(或)退出造成的样本量损失。

# 4.技术路线图



# 六、观察项目与检测时点

# 1.主要观察终点

以安全性作为研究的主要评价指标,包括单次 CART 输注后的 28 天和 3 个月剂量限制毒性(Dose-Limiting Toxicity, DLT)的类型 和发生率,以及 12 个月内 AE 的类型和发生率。

- (1) 剂量限制性毒性 (DLT)
- ① 定义。本研究中评价的 DLT 分别为两个时间窗,即发生在 CAR-T 细胞输注后的 28 天(第 0 天到第 28 天)和 3 个月(第 28 天 到第 3 个月)。该时间段的选择是基于 CAR-T 细胞在体内扩增、发挥活性和可能引起主要毒性的典型时间。

DLT 的判定必须满足以下全部条件:

- DLT 必须被研究者判定为很可能或肯定与CAR-T细胞输注相 关的不良事件,不能归因于基础疾病、合并症或伴随用药的毒 性;
- 不良事件必须达到≥3级严重程度等级(CTCAE标准 v5.0) 或≥3级特定毒性分级标准(如 IEC-HS 分级);
- ② 对于在 28 天和 3 个月内的 AE, 若符合以下任一条件将被定义为 DLT:
  - 无法控制的 3 级或≥4 级的 CRS;
  - 无法控制的 3 级或≥4 级的 ICANS;
  - 任何级别的 CRS 或 ICANS 导致死亡;
  - 任何≥3 级的非血液学毒性,包括但不限于: 3 级或以上的心脏 毒性(心肌炎、心衰)、肺毒性(急性呼吸窘迫综合征)、肝 毒性、肾毒性(急性肾损伤)、过敏反应等;
  - 持续性的≥4 级血细胞减少超过 28 天,排除了疾病进展或骨髓侵犯等其他原因。例如:白细胞(WBC)<1.0×10<sup>9</sup>/L;中性粒细胞(NEU)<0.5×10<sup>9</sup>/L等;

- 与 CAR-T 治疗相关的任何导致死亡的不良事件;
- 任何 CAR-T 相关且无法在 28 天内消退或控制的≥3 级毒性;
- 任何其他研究者或申办方认为具有临床意义并在未来足以限制剂量递增的严重毒性。
- ③ 对于研究中预期发生且易于管理的毒性(即使达到3级或以上)将不被定义为 DLT,排除的毒性事件包括:
  - 可控制的 3 级 CRS: 经标准支持治疗(托珠单抗和/或皮质类固醇)能在 72 小时内有效控制并降至<2 级:
  - 可控制的 3 级 ICANS: 经标准支持治疗(皮质类固醇)能在 72 小时内有效控制并降至≤2 级;
  - 短暂且易于管理的实验室异常,经过治疗后能在 28 天内恢复或有效控制并降至<2 级,如短暂性 3 级血细胞减少等。
    - (2) 不良事件(AE)

参考严重程度根据《不良事件通用术语标准》(CTCAE)V5.0) 进行分级:

- 1级: 轻度; 无症状或轻微; 仅为临床或诊断所见; 无需治疗。
- 2级:中度;需要较小,局部或非侵入性治疗;与年龄相当的工具性日常生活活动受限。
- 3级:严重或者具有重要医学意义但不会立即危及生命;导致住院或者延长住院时间;致残;自理性日常生活活动受限。
  - 4级: 危及生命; 需要紧急治疗。
  - 5级:与并发症相关导致的死亡。

# 2.次要观察终点

次要观察终点为有效性评价,包括 rMN 完全缓解(CR)、部分缓解(PR)、不缓解(NR)或复发情况:细胞输注后维持 CR、PR 的受试者比例、缓解的持续时间以及复发;和肾功能、免疫特征及细胞动态变化:蛋白尿、eGFR、血清抗 PLA2R 抗体、感染指标、补体、免疫球蛋白、细胞因子水平变化、血细胞、外周血免疫细胞亚群变化,CD19 在外周血 B 细胞亚群表面的表达水平等。

# (1) rMN 缓解或复发情况

细胞输注后 rMN 维持缓解、部分缓解或无缓解的受试者比例, rMN 缓解的持续时间以及 rMN 的复发。

- ① rMN CR 的定义。患者临床症状及体征消失,尿蛋白降至<0.3 g/d 或 UACR 为<300 mg/g,同时血清白蛋白(ALB)和血肌酐(Scr)水平正常;
- ② rMN PR 的定义。临床症状及体征好转,尿蛋白较基线下降超过50%,且尿蛋白降低至0.3~3.5g/d或UACR为300~3500 mg/g;
- ③ rMN 免疫学缓解的定义。PLA2R 抗体滴度低于 ELISA 检测阈值(2RU/mL)或间接免疫荧光试验结果为阴性;
- ④ rMN NR 的定义。蛋白尿下降不足或仍高,或肾功能恶化,不符合以上缓解、部分缓解或免疫学缓解的标准;
- ⑤ rMN 复发的定义。NR 或 PR 后,患者尿蛋白再次上升至>3.5 g/d 或 UACR>3500 mg/g;若复发次数在6个月内超过2次及以上或12个月内超过4次及以上,为频繁复发。

# (2) 肾功能、免疫特征及细胞动态变化

研究期间受试者血清尿素(BUN)、Scr、胱抑素 C (CysC)、eGFR、尿蛋白、UACR、血清抗 PLA2R 抗体、补体、免疫球蛋白、细胞因子水平变化、血细胞、CRP、CAR 拷贝参数、外周血免疫细胞亚群变化、CD19 在外周血 B 细胞亚群表面的表达水平等变化。

# (3) 检测时点

研究期间主要终点与次要终点的检测时点分别由表 3、4 所示。

| 结果测量 | 测度说明 | 时间框架 |
|--------------------|---------------------------|----------------|
| rMN 受试者单次输注 CD19 | | |
| CAR-T 细胞后 DLT 的类型和 | 参考研究方案中 DLT 定义 | 输注后 28 天和 3 个月 |
| 发生率 | | |
| rMN 受试者单次输注 CD19 | <br> 严重程度根据 CTCAE V5.0 进 | |
| CAR-T 细胞后 AE 的类型和发 | 行外级 | 输注后 12 个月 |
| 生率 | 11万级 | |

表 3. 研究主要终点(安全性)检测时点

| 表 4 | 研究次要终点 | (右泑性) | 粉测时占 |
|-------|--------|---------|------------------|
| AX 4. | 加力从安终总 | しつ ないまし | - 400 AVILLI II. |

| 结果测量 | 测度说明 | 时间框架 |
|---|---|---|
| 对于 rMN 受试者细胞输注后<br>的总缓解比例 | CR+PR | 输注后第2周、第1个月、第<br>2个月、第3个月、第6个月、<br>第9个月、第12个月、第18<br>个月(如适用)、第24个月<br>(如适用) |
| 对于 rMN 受试者细胞输注后<br>达到 CR 的比例 | 参照方案 CR 定义 | 输注后第2周、第1个月、第<br>2个月、第3个月、第6个月、<br>第9个月、第12个月、第18<br>个月(如适用)、第24个月<br>(如适用) |
| 对于 rMN 受试者细胞输注后<br>达到 PR 的比例 | 参照方案 PR 定义 | 输注后第 2 周、第 1 个月、第 2 个月、第 3 个月、第 6 个月、第 9 个月、第 12 个月、第 18 个月(如适用)、第 24 个月(如适用) |
| 对于 rMN 受试者细胞输注后<br>疾病复发的比例、频次及时 | 参照方案复发定义 | 输注后第2周、第1个月、第<br>2个月、第3个月、第6个月、 |

| 间 | | 第9个月、第12个月、第18 |
|---|---|---|
| 1~ | | 个月(如适用)、第24个月 |
| | | (如适用) |
| | | 输注后第2周、第1个月、第 |
| rMN 受试者单次输注 CD19 | | 2个月、第3个月、第6个月、 |
| CAR-T 细胞后 eGFR 与基线相 | 估计肾小球滤过率,采用 | 第 9 个月、第 12 个月、第 18 |
| 比的变化 | CKD-EPI2021 公式计算 | 个月(如适用)、第24个月 |
| MIJZI | | (如适用) |
| | | 输注后第2周、第1个月、第 |
| rMN 受试者单次输注 CD19 | | 2个月、第3个月、第6个月、 |
| CAR-T 细胞后尿蛋白与基线 | 24 尿蛋白定量 | 第 9 个月、第 12 个月、第 18 |
| 相比的变化 | » <b>(.</b> A A / C L | 个月(如适用)、第24个月 |
| | | (如适用) |
| | | 输注后第2周、第1个月、第 |
| rMN 受试者单次输注 CD19 | | 2个月、第3个月、第6个月、 |
| CAR-T 细胞后 UACR 与基线相 | 随机尿 | 第 9 个月、第 12 个月、第 18 |
| 比的变化 | | 个月(如适用)、第24个月 |
| | | (如适用) |
| | | 输注后第2周、第1个月、第 |
| rMN 受试者单次输注 CD19 | | 2个月、第3个月、第6个月、 |
| CAR-T 细胞后血清抗 PLA2R | 静脉血 | 第9个月、第12个月、第18 |
| 抗体与基线相比的变化 | | 个月(如适用)、第24个月 |
| | | (如适用) |
| | | 输注后第2周、第1个月、第 |
| rMN 受试者单次输注 CD19 | | 2个月、第3个月、第6个月、 |
| CAR-T 细胞后血清肾脏功能 | 静脉血, Scr、CysC | 第 9 个月、第 12 个月、第 18 |
| 与基线相比的变化 | | 个月(如适用)、第24个月 |
| | | (如适用) |
| | | 输注后第2周、第1个月、第 |
| rMN 受试者单次输注 CD19 | | 2个月、第3个月、第6个月、 |
| CAR-T 细胞后血细胞的变化 | 静脉血,血常规 | 第9个月、第12个月、第18 |
| | | 个月(如适用)、第24个月 |
| | | (如适用) |
| rMN 受试者单次输注 CD19 | \$-22. ∐ <del>``</del> | 输注后第2天、第7天、第 |
| CAR-T 细胞后 CRP 的变化 | 静脉血 | 10 或 14 天、第 21 天、第 28 |
| | | 天(1个月) |
| | | 输注后第2周、第1个月、第<br>2个月、第3个月、第6个月、 |
| rMN 受试者单次输注 CD19 | 血清补体 C3、C4 | 第 9 个月、第 12 个月、第 18 |
| CAR-T 细胞后补体的变化 | 111.4日本に入事でつい でも | 第9年月、第12年月、第18 <br> 个月(如适用)、第24 个月 |
| | | (如适用)、第24个月 |
| rMN 受试者单次输注 CD19 | | 输注后第2周、第1个月、第 |
| CAR-T 细胞后免疫球蛋白的 | IgE、IgA、IgG、IgM | 2个月、第3个月、第6个月、 |
| 变化 细胞/ 免疫坏蛋白的 | TEL TEU, TEU, TEM | 第 9 个月、第 12 个月、第 18 |
| Хru | | M 0 11 M 12 17 M 10 |

| | | 个月(如适用)、第 24 个月<br>(如适用) |
|---|---|---|
| rMN 受试者单次输注 CD19<br>CAR-T 细胞后 CAR 拷贝参数<br>的变化 | 与 CAR 拷贝数相关的参数 | 输注后第2天、第5天、第7<br>天、第10或14天、第21天、<br>第28天(1个月)、第2个<br>月、第3个月、第6个月、第<br>9个月、第12个月、第18个<br>月(如适用)、第24个月(如<br>适用) |
| rMN 受试者单次输注 CD19<br>CAR-T 细胞后铁蛋白的变化 | 铁蛋白水平 | 输注后第2天、第7天、10<br>或14天、第21天、第28天<br>(1个月) |
| rMN 受试者单次输注 CD19<br>CAR-T 细胞后细胞因子的变<br>化 | 细胞因子系列 | 输注后第2天、第7天、10<br>或14天、第21天、第28天<br>(1个月) |
| rMN 受试者单次输注 CD19<br>CAR-T 细胞后外周血淋巴细<br>胞亚群的变化 | 外周血淋巴细胞亚群计数 | 输注后第2天、第5天、第7<br>天、第10或14天、第21天、<br>第28天(1个月) |
| rMN 受试者单次输注 CD19<br>CAR-T 细胞后 CD19 在外周血<br>B 细胞亚群表面的表达水平 | 使用流式细胞仪方法 | 输注后第2天、第5天、第7<br>天、第10或14天、第21天、<br>第28天(1个月) |

# 七、不良事件的观察与处理

# (一) 淋巴细胞清除期

CAR-T 细胞回输前需要进行淋巴细胞清除预处理(以下简称清淋)为 CAR-T 细胞创造有利的免疫环境,改善其扩增、持久性和临床活性,同时降低抗 CAR 免疫应答。清淋潜在并发症包括全血细胞减少、免疫抑制、感染、出血性膀胱炎、肝肾损伤等,期间将每天监测受试者生命体征,24h 出入量,每 1~2 天监测全血细胞计数、肝肾功能等。

# (二) CAR-T 细胞回输后

CAR-T细胞回输后,患者需要接受密切的临床监测,以评估治疗的疗效和安全性。CAR-T细胞治疗的常见不良反应包括 CRS、ICANS、肿瘤释放综合征(TLS)、血细胞性淋巴组织细胞增生症/巨噬细胞活化综合征(HLHMAS)、CARAC、ICAHT、B细胞缺乏和低免

疫球蛋白血症、感染、过敏反应和 CAR-T 异常增殖等。本研究参考中国临床肿瘤学会(CSCO)CAR-T 细胞治疗恶性血液病指南(2024 年版)和中国嵌合抗原受体 T 细胞治疗难治性神经系统自身免疫性疾病专家共识(2025 年版),评估研究期间潜在的 CAR-T 细胞治疗相关的 DLT 及 AE,并制定相应的临床预防和处置预案。

# 1. 细胞因子释放综合征(CRS)

如果出现以下 4 种症状或体征之一,即应考虑 CRS 可能: (1) 发热,体温≥38℃; (2)低血压,收缩压<90 mmHg(1 mmHg=0.133 kPa); (3)动脉血氧饱和度<90%; (4)出现器官毒性。具体分级 参考美国移植和细胞治疗学会 CRS 分级方法<sup>[21]</sup>。

| 参数 | 1 级 | 2 级 | 3 级 | 4级 |
|---|---|---|---|---|
| 发热 | 体温≥38℃ | 体温≥38℃ | 体温≥38℃ | 体温≥38℃ |
| 低血压 | 无 | 有,不需要升压<br>药 | 需要升压药物<br>士 血管升压素 | 需要多种升压<br>药物(除外血管<br>升压素) |
| 低氧血症 | 无 | 有,需要低流量<br>鼻导管吸氧 | 需要高流量鼻<br>导管、面罩或文<br>丘里面罩吸氧 | 需要正压通气<br>(如 CPAP、<br>BiPAP、插管或<br>机械通气) |

表 5. CRS 的分级

注: CRS 相关的器官毒性可根据 CTCAE V5.0 进行分级,但不影响 CRS 分级; 发热的定义为体温≥38℃,且不属于任何其他原因。CRS 患者接受解热或使用珠 单抗或类固醇等抗细胞因子治疗,则后续 CRS 严重程度分级不再需要发热;低流 量鼻导管吸氧:≤6L/min:高流量鼻导管吸氧:>6L/min。

表 6. CRS 的处置措施

| 分级 | 症状或体征 | 处理 |
|---|---|---|
| 1级 | 发热(体温<br>≥38℃) | <ul><li>补充液体</li><li>对症降温:物理降温,对乙酰氨基酚或布洛芬等药物降温</li><li>排除感染:血尿培养、胸部影像学检查等</li><li>如患者存在粒细胞缺乏症,给予预防性应用抗生素,可</li></ul> |

| | | 使用 G-CSF,禁用 GM-CSF |
|----|--------------|----------------------------------------------------|
| | | • 如果持续发热(>3 天)或难治性发热,可予托珠单抗 |
| | | (8mg/kg),症状无改善者,可8小时后重复使用(建议 |
| | | 不超过3次) |
| | | • 治疗 24 小时后 CRS 无改善者,可予地塞米松 5~10mg qd |
| | | 或升级至2级处理 |
| | | • 补液、抗感染 |
| | | • 如果未使用过托珠单抗,可予托珠单抗(用法同1级) |
| | 医五尺子属 | • 1~2 剂托珠单抗治疗 CRS 无改善者, 予地塞米松 10mg q12h |
| 2级 | 低血压或低 | 或 qd,1~3 天,症状改善后尽快减量 |
| | 氧血症 | • 地塞米松处理 24 小时后无改善,按照 3 级处理 |
| | | • 低流量吸氧(如需要) |
| | | • 抗感染治疗 |
| | | • 考虑转入 ICU |
| | | • 补液、强效抗感染 |
| | 低血压或低<br>氧血症 | <ul><li>升压药物(如需要)</li></ul> |
| 3级 | | • 如果既往未使用过托珠单抗,可予托珠单抗(8mg/kg), |
| | | 用法同1级 |
| | | • 地塞米松 10~20mg q. 6h. ,1~3 天,症状改善后尽快减量 |
| | | <ul><li>高流量吸氧(如需要)</li></ul> |
| | | • 转入 ICU |
| | | • 高流量给氧或机械通气 |
| | | <ul><li>补液、强效抗感染</li></ul> |
| | 低血压或低 | <ul><li>多药升压(如需要)</li></ul> |
| 4级 | 氧血症 | ・ 大剂量糖皮质激素治疗(如甲泼尼龙 1g/d×3 天,逐步 |
| | 半、川川川に | 一人的重幅反应做系和为(如于极地况 1g/u/3 八,逐少 <br> 減量 ) |
| | | 〜<br> ・<br> ・<br> ・<br> ・<br> ・<br> ・<br> ・ |
| | | • 持续监测和支持治疗 |

注:托珠单抗单次治疗最大剂量为800mg,可重复给药。治疗后24小时CRS 无改善甚至加重,应升级至下一级处置措施。托珠单抗和类固醇的早期干预不会 影响体内CD19 CAR-T细胞的扩增和疗效。

# 2. 免疫效应细胞相关神经毒性综合征(ICANS)

ICANS 临床表现多样,早期症状常表现为注意力减弱、语言障碍、书写能力减退等,其中测试书写能力是评估 ICANS 进展的一种相对简单且敏感的衡量方法。大多数患者 ICANS 临床症状呈可逆性,少数患者可出现严重的临床症状,表现为癫痫发作、精神错乱、颅内压增高等。最严重可进展为急性脑水肿,患者可在数小时内从轻度的

嗜睡进展为意识不清,进一步发展导致死亡。具体分级参考美国移植和细胞治疗学会 ICANS 分级方法<sup>[21]</sup>。

ICANS 的症状和体征通常在 CAR-T 细胞回输后第 3~6 天出现,第 7~8 天达到高峰,后随着时间推移而逐渐改善,持续 2~3 周症状消失<sup>[22]</sup>。本研究中除密切监测患者血常规、血生化、凝血功能、铁蛋白、细胞因子水平等指标,一旦研究者或临床医生怀疑 ICANS,在排除禁忌症后,根据受试者情况将进行脑脊液检查、头颅 CT/MRI 和脑电图检查。

| 参数 | 1级 | 2级 | 3 级 | 4 级 |
|---|---|---|---|---|
| ICE 评 | 7-9 | 3-6 | 0-2 | 0(患者不能唤醒,无法进行 |
| 分*/分 | 1 9 | 3 0 | 0 2 | ICE 评分) |
| 意识下 | 自然 | 声音 | <br> 仅可通过触觉刺激唤醒 | 不能唤醒或需强烈/反复刺 |
| 降 <sup>†</sup> | 唤醒 | 唤醒 | | 激; 昏迷 |
| 癫痫‡ | N/A | N/A | 可快速缓解的局部/全<br>身癫痫发作;或干预后<br>缓解的非惊厥性癫痫<br>(脑电图) | 持续癫痫(>5 分钟)或反复<br>发作无法恢复基线 |
| 运动障 碍 | N/A | N/A | N/A | 深度局部运动减弱(如偏瘫、<br>轻瘫) |
| 颅内压<br>增高/<br>脑水肿 <sup>§</sup> | N/A | N/A | 神经影像学发现局灶/<br>局部水肿 | 弥漫性脑水肿;去脑/去皮质<br>状态;脑神经VI麻痹;视神<br>经盘水肿;库欣三联征 |

表 7. ICANS 的分级

注: ICANS 分级由不属于任何其他原因的最严重事件确定。应考虑基线 ICE 水平在输注 CAR-T 之前评分。

\*免疫效应细胞相关脑病(ICE)评分为 0 分的患者如果清醒时有完全性失语 归类为 3 级 ICANS,但 ICE评分为 0 分的患者如果无法唤醒,则被归类为 4 级 ICANS。 具体评分细则:定向(4分):年,月,城市,医院;命名(3分):3个物体(如时钟、 笔、纽扣);遵循指令(1分):如伸出两个手指、闭眼和伸舌;书写(1分):能够写 标准语句(如"我们的国旗是五星红旗");注意力(1分):从 100 每隔 10 个数倒数。

- +没有其他原因(如没有使用镇静药物)。
- ‡与免疫效应细胞治疗相关的震颤和肌阵挛可根据 CTCAEV5. 0 进行分级,但它们没有影响评分。

§颅内出血或脑梗死伴或不伴水肿不被认为是神经毒性特征,并被排除在ICANS 分级之外。它可根据 CTCAE V5.0 进行分级。

表 8. ICANS 的处置措施

| 分级 | 推荐处理方法 |
|------|-----------------------------------------------|
| | • 吞咽功能受影响时: 口服药物及营养改为静脉输注 |
| | • 躁动患者: 低剂量劳拉西泮或氟哌啶醇镇静 |
| | • 神经科会诊 |
| | • 眼底镜检查(评估视神经盘水肿) |
| | • 颅脑影像学检查(增强 MRI/CT) |
| 1级 | • 可选腰穿(检测颅内压、细胞因子、CAR-T 细胞数) |
| 1 30 | • 脑电图检查 |
| | • 预防性处理: |
| | - 地塞米松 5-10mg (若可能进展为严重神经毒性) |
| | - 左乙拉西坦(预防癫痫) |
| | • 合并 CRS 时:托珠单抗 8mg/kg (未使用过抗 IL-6 治疗者),8 小时后 |
| | 可重复(总量≤2-3 次) |
| | • 同1级对症处理及检查 |
| | • 合并 CRS 时: 托珠单抗用法同 1 级 |
| | • 抗 IL-6 无效或未合并 CRS 时: |
| 2级 | - 地塞米松 10mg q6-12h 或 |
| | - 甲泼尼龙 1mg/kg q12h (症状降至1级后快速减量) |
| | • 合并≥2 级 CRS: 建议转入 ICU |
| | • 影像学检查: 每 2-3 天重复 |
| | • 同1级对症处理及检查 |
| | • 立即转入 ICU, 机械通气支持 |
| | • 大剂量激素治疗: |
| 3级 | - 甲泼尼龙 1g/d×3 天 → 逐步减量(250mg q12h×2 天 → 125mg |
| | q12h×2 天 → 60mg q12h×2 天) |
| | • 抗 IL-6 治疗原则同 3 级 |
| | • 糖皮质激素无应答时: 考虑阿那白滞素(IL-1 受体拮抗剂) |

注:由于托珠单抗与 IL-6 受体结合后导致血清游离儿-6 水平升高,进一步增加脑脊液中 IL-6 浓度,有可能加重神经毒性。在 ICANS 的处理过程中,糖皮质激素的使用较托珠单抗更重要。

# 3. 免疫效应细胞相关噬血细胞性淋巴组织细胞增生症样综合征 (IEC-HS)

IEC-HS 是一种独立于 CRS 和 ICANS 的病理和生化过度炎症反应综合征,具有以下特点:

- (1)表现为巨噬细胞活化(MAS)/血细胞淋巴组织细胞增生(HLH)的特征:
  - (2)归因于免疫效应细胞治疗;
- (3)加重或新发的血细胞减少症、高铁蛋白血症、伴有低纤维蛋白原血症的凝血异常和/或转氨酶异常。除此之外,IEC-HS通常被认为是 CRS 处理过程后的延迟表现。

IEC-HS 定义为基于免疫效应细胞治疗后出现的病理和生化高炎症状态的综合征,具体为巨噬细胞活化综合征(MAS)或噬血细胞性淋巴组织细胞增多症(HLH)。IEC-HS 的发生独立于 CRS 和 ICANS,伴随血细胞减少、高铁蛋白血症、凝血功能障碍伴低纤维蛋白原血症、转氨酶升高等的新发或加重。除此之外,IEC-HS 通常被认为是 CRS 处理过程后的延迟表现。

#### 表 9. IEC-HS 的诊断标准\*

# ・ 铁蛋白升高(>2×ULN 或输注时基线)和/或快速升高(临床评估) ・ CRS 治疗初步改善或消退后炎症反应加重 ・ 肝转氨酶升高(>5×ULN (基线正常) <sup>6</sup>或>5×基线值(基线异常) <sup>‡</sup> ・ 低纤维蛋白原血症(<150mg/d1 或<LLN) <sup>#</sup> ・ 骨髓或其他组织中噬血现象<sup>#</sup> ・ 不以上的 4 级血细胞减少症(新发、加重或难治性) <sup>&</sup> ・ 乳酸脱氢酶升高(>ULN) ・ 凝血异常(如 PT/APTT 升高) ・ 高直接胆红素血症 ・ 新发脾肿大 ・ 发热(新发\*或持续\*)

- 中枢神经系统毒性
- 肺部表现(缺氧、肺部浸润、肺水肿)
- 新发肾功能不全
- 高甘油三酯血症(空腹>265mg/d1)#

注: ULN:正常值上限; LLN:正常值下限。

\*仅在不能归因于其他病因(包括 CRS、感染和/或疾病进展)的情况下做出诊断。

†指同时出现的症状群(如所有症状都在72小时内出现)。

‡虽然大多数 IEC-HS 病例都有 CRS, 但并不绝对。

§符合 CTCAEV5.0 中的3级转氨酶升高

#参考 HLH-2004。

&通常指血象至少一系出现 4 级血细胞减少(血小板、中性粒细胞、血红蛋白)。 ※与 CRS 初发或复发鉴别。

#### 表 10. IEC-HS 的分级

| 分级 | 症状严重程度和干预措施 |
|-------|---------------------------------|
| | 无症状或轻微症状 |
| 1级 | • 仅需观察和临床评估 |
| | • 持续临床监测 |
| | 轻度至中度症状 |
| 2级 | • 需医疗干预(如: |
| 2级 | - 免疫抑制剂治疗(针对 IEC-HS) |
| | - 无症状低纤维蛋白原血症的输血支持) |
| | 严重症状(非即刻危及生命) |
| 2 414 | • 需积极治疗(如: |
| 3级 | - 输血支持的出血性凝血功能障碍 |
| | - 因新发急性肾损伤/低血压/呼吸窘迫需住院) |
| A GTG | 危及生命的症状需紧急干预(如:危及生命的出血或低血压、需插管的 |
| 4级 | 呼吸窘迫或需透析的急性肾损伤) |
| 5 级 | 死亡 |

#### 表 11. IEC-HS 的处置措施

| 治疗<br>级别 | 推荐方案 |
|----------|--------------------------------------------------------|
| 一级 | <ul><li>阿那白滞素(200-800mg/天)</li><li>和/或糖皮质激素:</li></ul> |
| 治疗 | - 地塞米松 10-40mg/天 |
| 二级 | - 或 甲泼尼龙 1000mg/天 • 48 小时未缓解时: |
| 治疗 | - 增加一线药物剂量 |

| | - 采用双联治疗(阿那白滞素+糖皮质激素) |
|----------|----------------------------------------|
| | - 可加用 JAK-2 抑制剂 (如芦可替尼 5-10mg/天) |
| | • 加用 JAK-2 抑制剂 |
| | • 可考虑: |
| 三级 | - γ干扰素单克隆抗体(依马利尤) |
| 治疗 | - CTLA-4 激动剂(如阿巴西普) |
| | - CD52 抗体 (阿仑单抗) |
| | • 依托泊苷(50-100mg/m²)适用于原发性 HLH 和继发性 HLH |
| 松米 | • 快速进展/危及生命的高级别 IEC-HS: |
| 挽救<br>治疗 | - 一/二线治疗失败后 |
| 144)1 | - 可考虑 TKI (如达沙替尼) 作为三线选择 |

注:由于缺乏前瞻性研究和 IEC-HS 治疗方法的数据,因此治疗考量来源于专家共识意见。共识中提到目前对于三线及后续治疗方案的选择较多,因此,若研究中出现 IEC-HS,研究者或临床医生将根据患者的具体情况采用相应的治疗方法。

表 12. IEC-HS 的支持性治疗

| 治疗<br>类型 | 推荐处理方法 |
|---|---|
| 监测 | <ul> <li>每日监测:</li> <li>血常规、凝血功能、纤维蛋白原</li> <li>肝肾功能异常患者的日常评估</li> <li>感染监测:</li> <li>血/尿/痰培养(细菌、病毒、真菌)</li> <li>其他感染源检测(如肺泡灌洗液、脑脊液)</li> <li>HLH 相关参数:</li> <li>可溶性 CD25、NK 细胞功能、甘油三酯</li> <li>骨髓涂片、IFN-γ、CXCL9/CXCL10、IL-10/IL-18</li> </ul> |
| 血细<br>胞减<br>少症 | <ul> <li>维持血红蛋白&gt;7g/d1</li> <li>维持血小板&gt;50×10°/L(活动性出血或凝血功能障碍时)</li> <li>ANC&lt;0.5×10°/L时可考虑G-CSF(存在争议)</li> <li>月经过多患者建议妇科诊治</li> </ul> |
| 凝血<br>功能<br>障碍 | <ul> <li>维持纤维蛋白原: <ul> <li>&gt;100mg/dl (无出血)</li> <li>&gt;150mg/dl (伴出血)</li> </ul> </li> <li>INR&gt;1.5 时补充维生素 K</li> <li>INR&gt;2 时给予冷沉淀和 FFP</li> <li>慎用静脉血栓栓塞预防药物</li> </ul> |
| 感染管理 | 经验性抗感染治疗 排除感染性 sHLH 病因 免疫抑制治疗期间需预防性抗感染 定期感染监测 |

# 4. CAR-T 相关出凝血性疾病(CARAC)

CRS 会引起患者出凝血功能障碍。处理原则为早期识别、准确评估、去除诱因、依据 CRS 分级进行分层干预。CARAC 的参考处理方法如下表。

表 13. CARAC 的处置措施

| CRS<br>分级 | CARAC 管理 | 预防和支<br>持治疗 | 预防/抗<br>感染治疗 | 抗炎和护<br>肝治疗 | 促血小板<br>生成 |
|---|---|---|---|---|---|
| 1级 | • 评估凝血指标: 若正常: 观察。若异常: ① 增加凝血指标监测频率 ② WHO 出血评分 ③ 密切监测 CRS | √<br>√ | √<br>√ | <i>√</i> | <i>✓</i> |
| 2级 | • 评估凝血指标: 若改善: 观察。<br>无改善: 观察。<br>无改善: ① 增加监测频率<br>② WHO 出血评分+DIC 评分<br>③ 控制 CRS(细胞因子拮抗剂+糖皮质激素)<br>④ 替代和抗凝治疗 | √ | √ | √ | √ |
| 3级 | • 评估凝血指标: 若改善: 观察。<br>无改善:<br>① 增加监测频率<br>② WHO 出血评分+DIC 评分<br>③ 加强 CRS 控制(增加糖皮质激素剂量/频率)<br>④ 以替代治疗为主<br>⑤ 适时调整方案 | ✓ | √ | √ | ✓ |
| 4级 | • 评估凝血指标: 若改善: 观察''<br>无改善:<br>① 增加监测频率<br>② WHO 出血评分+DIC 评分<br>分 | √ | √ | √ | <b>√</b> |

| 法联合) |
|-------------|
| ④ 替代治疗+血浆置换 |

# 5. 免疫效应细胞相关血液毒性(ICAHT)

部分患者可能会发生血细胞三系下降,持续半年甚至更久。应密 切关注血细胞下降期间感染风险的增加,必要时给予造血刺激因子, 输注血液制品如浓缩红细胞和血小板。

分级 Ι级 II 级 III 级 IV 级 早期 ICAHT≤30 天 ANC  $\leq$  500/  $\mu$  1 <7 天 从未> 500/μ1 >7-13 天 ≥14 天 ANC  $\leq 100/\mu 1$ ≥14 天 ≥7 天 晚期 ICAHT>30 天 ANC  $\leq 1 500/\mu 1$  $\checkmark$ ANC  $\leq$  1 000/  $\mu$  1  $\checkmark$ ANC  $\leq$  500/  $\mu$  1 ANC  $\leq 100/\mu 1$  $\checkmark$ 

表 14. ICAHT 分级标准

注: ANC, 中性粒细胞绝对值, 多次测量, 非一过性减少。

| 评估指标 | 0 分 | 1分 | 2 分 |
|---|---|---|---|
| 血小板计数 | $>175 \times 10^{9}/L$ | $75-175 \times 10^9 / L$ | $<75 \times 10^{9}/L$ |
| 中性粒细胞绝对值 | $>1.2 \times 10^9/L$ | $<1.2\times10^{9}/L$ | |
| 血红蛋白 | >90g/L | <90g/L | |
| C 反应蛋白 | <30mg/L | ≥30mg/L | |
| 铁蛋白 | <650ng/ml | 650-2,000ng/ml | >2,000ng/m1 |

表 15. CAR-HEMATOTOX 的风险分层评分

注: 低危 0-1 分, 高危>2 分, 根据清淋前(-5 天, 宽限期 3 天)结果评估血液毒性及感染发生率, 高危患者血液毒性及感染发生率明显增加。

| 表 16. | ICAHT 短期官均 | 里的处埋万法 |
|-------|------------|--------|

| 处理措施 | 时间 | 方式 | 注意事项 | 备注 |
|---|---|---|---|---|
| 浓缩红细胞<br>(pRBC)或血<br>小板输注 | 基于患者血细<br>胞下降风险特<br>征 | 对于 pRBC, 考虑每次使用 1个产品,以减少铁过载 | 血液制品辐照或滤除白细胞;从单采前7天开始,直到CAR-T后至少90天 | Flu 可能会影响辐照血液制品 |
| G-CSF 预防 | 具有 ICAHT 高 | G-CSF 5μg/kg | ICAHT 低危患 | 降低发热性粒 |
| 性使用 | 危特征患者在 | qd | 者可能不需要 | 细胞减少症风 |

| | <b>然</b> 。 | | 0.000 | 7/ / <del>7</del> 1×1> 0 |
|---|---|---|---|---|
| | 第+2 天预防使 | | G-CSF | 险(不增加≥3 |
| | 用 | | | 级 CRS 或 |
| | | | | ICANS 风险) |
| | | | | 中性粒细胞间 |
| G-CSF 治疗 | ANC<500/ μ 1 | 5μg/kg qd, | | 歇性恢复患者 |
| 性使用 | MNC SOO/ μ1 | 无应答时考虑 | _ | 反应迅速,再 |
| 正使用 | h.1 | 10 μ g/kg | | 生障碍性患者 |
| | | | | 无反应 |
| | | G-菌: 三代/四 | | 根据治疗期间 |
| | ANC<500/ μ 1 | 代头孢、酶复 | MRD、CRE 等病 | 医疗中心所在 |
| 细菌预防 | 时考虑预防治 | 合制剂; G+菌: | 原体定植时注 | 地及患者常住 |
| | 疗 | 万古霉素、替 | 意 | 地的细菌流行 |
| | | 考拉宁等 | | 病学调整 |
| | 从清淋预处理 | 伐 昔 洛 韦 | | |
| | 开始至 CAR-T | K 日 日 日 日 日 日 日 日 日 日 日 日 日 日 日 日 日 | | |
| 病毒预防 | 后1年和/或 | 阿普洛韦 | _ | _ |
| | $CD4^+ > 0.2 \times 1$ | 800mg bid | | |
| | 0°/L | Oooliig Did | | |
| | 从清淋预处理 | | | |
| │<br>│ 肺孢子虫预 | 开始至 CAR-T | 复方新诺明 | 过敏者可选用 | |
| 防 | 后1年和/或 | 480mg qd 或 | 喷他脒、氨苯 | _ |
| Line | $CD4^{+}>0.2\times10^{9}$ | 960mg tiw | 砜或阿托伐醌 | |
| | /L | | | |
| | 中性粒细胞减 | 泊 沙 康 唑 | 既往有侵袭性 | |
| 霉菌预防 | 中 E 松 细 胞 | 300mg/d 或米 | 曲霉病或长期 | _ |
| <b>每</b> 图 | | 卡芬净 500mg | 使用皮质类固 | _ |
| | 月 | i.v./d | 醇者建议预防 | |

注:基线血细胞减少症、发生>3级 CRS 或 ICANS、长期使用糖皮质激素、CAR-HEMATOTOX 评分为高危的受试者感染风险可能较高。

# 6. B细胞缺乏症/低丙种球蛋白血症

B细胞发育不全被定义为一种由B细胞耗竭或缺失引起的疾病。 CAR-T 诱导的B细胞发育不全的机制为靶向CD19的CAR-T的细胞疗法非肿瘤靶向毒性(On-target off-tumor efect)及脱靶毒性(Off-target effects),通常是因为靶点为共享靶点,在正常组织同样表达,会被CAR-T识别攻击,而引起的毒性。这一类毒副作用在CAR-T较为常见,其严重程度与靶点在正常组织的表达与作用关键程度相关,可降 低B细胞计数和丙种免疫球蛋白的水平。

目前,CAR-T临床报道的脱靶毒性案例并不多,可能原因是 CAR使用的单链抗体(scFv)多为高亲和力单抗,且很多抗体药物本身已经在临床上使用,证明安全性良好,从而保证了 CAR-T 的安全性。但是在 CAR-T 细胞回输后依旧需要注意其 Off-target effects,研究显示,CAR-T 回输后不同时间段均可能发生低丙种球蛋白血症,90 天后发生率约 67%,少数患者甚至持续数年。临床主要表现为频繁的感染。

(1) B细胞绝对值计算方法:B细胞绝对值=白细胞总数×淋巴细胞%x(CD19+或 CD20+)%,

定义/范围: B细胞绝对值<61 个细胞/ml; IgG≤400mg/dl。

- (2) 处理策略: 静脉滴注人免疫球蛋白(5g×3天,静脉滴注) 替代治疗。
- (3)输注频次: CAR-T 回输后 1 次/月,直至 B 细胞恢复至正常范围或 CAR-T 输注满 6 个月;高危人群持续 1 次/月,直至高危因素解除并且球蛋白水平恢复正常。针对 IgG≤400mg/dl 伴严重感染、持续感染或反复感染的高危人群,注意定期监测血清 IgG、IgM、IgA及外周血中(CD19+或 CD20+B 细胞数量等。

表 17. B 细胞缺乏症/低丙种球蛋白血症的分级和处理措施

| 分级 | 处理措施 |
|---|---|
| 任何级别 | <ul> <li>建议接种流感和 COVID-19 疫苗</li> <li>病毒预防和 PCP 预防(持续至 CAR-T 输注后 6-12 个月和/或 CD4 细胞计数&gt;200 个/μ1)</li> <li>高危患者*考虑抗真菌预防(如泊沙康唑),包括接受皮质类固醇治疗 CRS/ICANS 者</li> </ul> |
| 1级 | • 无需特殊干预 |

| (无症状) | • 对症支持治疗 |
|---------------------|-------------------------------------------------|
| 2级<br>(有症状,<br>非紧急) | |
| 3 级<br>(需紧急干<br>预) | • IgG≤400mg/dL 时考虑 IVIG 替代治疗<br>• 感染状态下针对性抗感染治疗 |
| 4 级<br>(危及生<br>命) | |

\*真菌感染高危标准(满足≥2 项): 输注前 ANC≤0.5×10°/L, CAR-T 剂量 >2×10<sup>7</sup>/kg

# 7. 感染

CAR-T细胞治疗后各种类型感染发生率约为 55%, 其中>3 级的严重感染约为 33%, 大部分感染发生在接受 CAR-T细胞治疗后 1~2年内, 其中 CAR-T细胞治疗后 1个月内感染发生率可高达 40%。CAR-T治疗后因感染部位不同,可出现发热、咳、咳痰、低血压等非特异性症状,严重时可导致血压下降、缺氧等系统性症状。感染风险增加与以下因素有关:既往治疗的次数、近 100 天内的感染、糖皮质激素或托珠单抗的使用、发热性中性粒细胞减少、靶向 CD22的CAR-T细胞疗法、低丙种球蛋白血症,早期严重感染的其他潜在危险因素包括 ICANS、托珠单抗和皮质类固醇使用。

# (1) 感染筛查

表 18. 受试者入组/接受 CAR-T 细胞回输前需要完成的感染筛查

| | 项目 |
|-------|---------------------------------------|
| 常规检查 | 病史询问和体格检查,感染性疾病(侵袭性真菌病、肝炎、梅毒、 |
| | 艾滋病、结核),其他重要的疾病史 |
| 实验室检查 | 血尿便常规、血沉、肝肾功能、电解质、免疫球蛋白、降钙素原、 |
| | C 反应蛋白、IL-6 等细胞因子检测(基线) |
| 病原学检查 | HCV、HBV、HIV、TP、EBV、CMV、新冠病毒检测,根据患者情况必 |
| | 要时增加 HSV/VZV、JCV、呼吸道相关病毒、支原体、G/GM 试验、 |

# (2) 感染预防

版本号:

感染发生高峰时期一般为 CAR-T 细胞输注后 8 周内,随时间延长而下降,可持续至治疗后 1~2 年。CRS 反应期合并感染的死亡率高,因此,感染防控是 CAR-T 细胞治疗的重中之重。

本研究期间受试者感染的管理主要参考《嵌合抗原受体 T 细胞治疗相关感染预防、诊断及治疗中国专家共识(2022 年版)》。清淋开始时给予阿昔洛韦或伐昔洛韦,用药时间根据免疫功能恢复情况确定。输注 CAR-T 细胞至粒细胞恢复前给予诺氟沙星、三唑类抗真菌药及复方磺胺甲恶唑片等预防感染(对于喹诺酮类、磺胺类药物等过敏的患者,可替换为青霉素类或头孢类、大环内酯类抗生素)。

表 19. CAR-T 治疗期间感染预防方案

| 感染类型 | 药物及剂量 | 用药时长 | 备注 |
|---|---|---|---|
| 细菌 | _ | _ | 目前尚无循证医学<br>证据支持在免疫治<br>疗同时予以常规细<br>菌预防 |
| 病毒* | <ul> <li>阿昔洛韦 400mg q12h 口服</li> <li>或 5mg/kg q12h 静脉注射</li> </ul> | 自清淋预处理开<br>始至 CAR-T 回输<br>后 6 个月; 高危<br>患者 <sup>†</sup> 延长至 1 年 | • 常规预防<br>• 高危患者加强监<br>测 |
| 侵袭性真菌 | <ul> <li>氟康唑 400mg qd</li> <li>丝状真菌预防:</li> <li>泊沙康唑 200mg tid p.o.<br/>(混悬剂)</li> <li>或 300mg qd p.o. (片剂,首日 bid)</li> <li>米卡芬净 50mg qd i.v.</li> </ul> | 直至中性粒细胞<br>恢复正常 | <ul><li>所有患者: 氟康唑预防</li><li>高危患者: 加用丝状真菌预防</li></ul> |
| 肺孢子虫 | <ul> <li>首选:复方新诺明<br/>(TMP/SMX 160/800mg) bid 2<br/>次/周</li> <li>替代:喷他脒 300mg 雾化</li> </ul> | 回输前1周开始<br>至 CD4 细胞计<br>数>200个/µ1 | 所有患者均需预防 |

毎月1次

\*CMV、EBV 监测: CMV、EBV 血清学 IgG+, IgM-患者,治疗期间应每 1~3 个月进行病毒 PCR 监测。慢性 HBV、HCV 感染患者与肝病专家共同管理,制定合理的管理流程。

†近期接受类固醇/托珠单抗治疗。

# (3) 感染处理

① 治疗期间感染的处置原则

表 20. CAR-T 治疗期间感染处置原则

| 分级 | 处理措施 |
|---|---|
| 任何级别 | <ul> <li>预防性抗病毒和肺孢子菌肺炎(持续至 CAR-T 输注后 6-12 个月和/或 CD4 细胞计数&gt;200 个/μ1)</li> <li>高风险患者考虑抗真菌预防</li> <li>CRS 后持续&gt;7d 中性粒细胞减少者可使用 G-CSF</li> </ul> |
| 1 级<br>(轻微感染) | <ul><li>支持治疗</li><li>发热时经验性抗感染:</li><li>抗细菌:如左氧氟沙星/环丙沙星</li><li>抗真菌:如氟康唑</li><li>抗病毒:如伐昔洛韦/阿昔洛韦</li></ul> |
| 2级<br>(需口服抗<br>生素) | • 按疗程口服抗菌药物 |
| 3级(严重感染) | <ul><li>静脉使用抗菌药物</li><li>全身性抗感染治疗</li></ul> |
| 4 级<br>(危及生命) | • 重症监护支持 |

# ② 治疗期间特殊状态下感染的管理

# a. CRS 与感染鉴别

两者临床表现有相似之处,但目前尚无特异性的标志物将两者明确区分开来,且 CRS 合并感染的情况可能发生,因此,对两者的发生发展的预判及干预时机把握至关重要。CRS 分级与感染程度在细胞因子水平上并未显示出明显的差异。当 CRS 合并严重感染时,可能会出现 IL-6 水平的二次升高,可尝试通过 II-8、IL-1 β、IFN 等细胞

因子来鉴别 CRS 与感染,但目前仍缺乏足够的临床数据与证据。若两者无法明确鉴别,以预防性抗感染联合 CRS 分级治疗为指导原则。

#### b. 特殊感染监测

包括结核、组织胞浆菌病、李斯特菌病和诺卡菌病等。研究者和 临床医生应注意病史询问,特别是在常规抗感染药物治疗无效时,需 考虑此类特殊病原菌感染可能。

# c. 确诊新型冠状病毒感染患者

患者自招募入组至 CAR-T 细胞回输期间出现新冠病毒感染时,应推迟 CAR-T 细胞治疗。对于无症状患者,CAR-T 回输应自首次核酸检测阳性之日起推迟≥14 天;对于轻度症状患者,CAR-T 回输应自症状好转,并且在不使用退热药物的情况下退热至少 24 小时后起算,推迟≥14 天。若患者持续性核酸检测阳性或症状未缓解或进行性加重,经研究团队评估后,应退出本研究。

# 8. 过敏反应

通常发生于细胞输注后 2 周内的皮疹,表现为压之褪色,3~5d 可自行消退,发生原因除过敏外,可能为细胞因子释放导致毛细血管内皮脆性增加,伴或不伴有血小板减少,需结合多项指标综合评判。药物过敏的原因可能来自 CAR-T 生产过程中的体外培养试剂成分、病毒载体杂质、CAR-T 前未恢复的炎性背景导致的 T 细胞活化等。

本研究期间对于 CAR-T 相关过敏反应的管理措施主要包括:入 组时排除有超敏或过敏反应的患者,在 CART 细胞制造过程中严格控 制程序和试剂,预防性使用抗过敏药物(如苯海拉明或异丙嗪等)、 CAR-T细胞回输后 14d 内密切监测患者生命体征及症状。

# 9. CAR-T细胞异常增殖

CAR-T细胞回输 28d 内,监测外周血 CAR-T细胞体内扩增,前 1周内每 2~3 天采集 1次血样此后每周采集 1次。具体时间点为:输注后第 2 天、第 5 天、第 7 天、第 10 或 14 天、第 21 天、第 28 天。

CAR-T 细胞异常增殖诊断标准为: 外周血白细胞计数>10×10<sup>9</sup>/L; 白细胞中淋巴细胞百分比≥70%; CAR-T 细胞绝对计数>600 个/μl。

当考虑患者出现 CAR-T 细胞异常增殖时,予以糖皮质激素和其他免疫抑制剂(例如抗胸腺细胞球蛋白或抗 CD52 抗体)。病情严重的患者可联合使用 2 种或 2 种以上免疫抑制剂。

# 八、研究的质量控制与质量保证

研究者将负责遵照纳入排除标准筛选受试者,在 CRF 中记录研究数据,并将研究数据输入电子数据库中。同时,严格按照时间节点,保持与受试的密切联系。避免入选不合格的研究对象、研究的受试者自动退出、受试者根本没有接受治疗等现象的发生。由专人独立进行研究监测、数据管理、安全监测和统计分析。一旦完成质量保证程序,数据库将被锁定。

# 九、统计学处理

所有统计分析都不考虑受试者依从性差、中途退出或失访等情况。由于本研究样本量较小,所有数据均以个体数值呈现。研究将采用描述性统计方法报告基线期和随访期的特定参数,统计分析和数据展示使用 SPSS 27.0 和 GraphPad Prism9.0 版本完成。

基线特征按个体 ID 逐例列出:包括年龄、性别、病理分型、基线尿蛋白、抗 PLA2R 抗体水平等。

连续变量的变化如实验室指标,按照受试者个体 ID 记录个体随 访数值表格,和/或绘制多时间点折线图(时间轴图谱[从输注日至 D+n 天])。分类变量 ,按照个体状态标注(例: CR/PR/NR)。安全性事件按个体列出毒性类型、分级、发生时间、持续时间、干预措施、转归等。

因样本量仅5例,所有发现均为描述性,不代表总体推断。

# 十、临床研究的伦理学

临床研究将遵循世界医学大会《赫尔辛基宣言》等相关规定。在研究开始之前,由伦理委员会批准该试验方案后方可实施临床研究。每一位受试者入选本研究前,研究者有责任向受试者或其法定代理人完整、全面地介绍本研究的目的、程序和可能的受益及风险,并签署书面知情同意书,应让受试者了解他们有权随时退出本研究,知情同意书应作为临床研究文件保留备查。研究过程中将保护受试者的个人隐私与数据机密性。

# 十一、研究进度

2025年08月01日-2025年10月31日:前期准备,研究方案设计, 召开研究者会议,伦理委员会审核、试验注册。

2025年11月01日-2026年03月31日: 试验启动,患者入组随访, 监察员访视,数据收集、血液标本、药物不良事件的管理。 2026年04月01日-2028年7月31日: 数据汇总,资料保存,统计

# 分析处理,撰写并发表论文,报告结果。

# 十二、参考文献

- [1] DANTAS M, SILVA L B B, PONTES B T M, et al. Membranous nephropathy [J]. Jornal brasileiro de nefrologia, 2023, 45(2): 229-43.
- [2] KERI K C, BLUMENTHAL S, KULKARNI V, et al. Primary membranous nephropathy: comprehensive review and historical perspective [J]. Postgrad Med J, 2019, 95(1119): 23-31.
- [3] HOU J H, ZHU H X, ZHOU M L, et al. Changes in the Spectrum of Kidney Diseases: An Analysis of 40,759 Biopsy-Proven Cases from 2003 to 2014 in China [J]. Kidney diseases (Basel, Switzerland), 2018, 4(1): 10-9.
- [4] WANG M, YANG J, FANG X, et al. Membranous nephropathy: pathogenesis and treatments [J]. MedComm (2020), 2024, 5(7): e614.
- [5] SETHI S, BECK L H, JR., GLASSOCK R J, et al. Mayo Clinic Consensus Report on Membranous Nephropathy: Proposal for a Novel Classification [J]. Mayo Clin Proc, 2023, 98(11): 1671-84.
- [6] ALSHARHAN L, BECK L H, JR. Membranous Nephropathy: Core Curriculum 2021 [J]. American journal of kidney diseases: the official journal of the National Kidney Foundation, 2021, 77(3): 440-53.
- [7] DENG L, XU G. Update on the Application of Monoclonal Antibody Therapy in Primary Membranous Nephropathy [J]. Drugs, 2023, 83(6): 507-30.
- [8] ROJAS-RIVERA J, FERVENZA F C, ORTIZ A. Recent Clinical Trials Insights into the Treatment of Primary Membranous Nephropathy [J]. Drugs, 2022, 82(2): 109-32.
- [9] FERVENZA F C, APPEL G B, BARBOUR S J, et al. Rituximab or Cyclosporine in the Treatment of Membranous Nephropathy [J]. N Engl J Med, 2019, 381(1): 36-46.
- [10] GAUCKLER P, SHIN J I, ALBERICI F, et al. Rituximab in Membranous Nephropathy [J]. Kidney Int Rep, 2021, 6(4): 881-93.
- [11] KITCHING A R, JAW J. Chimeric antigen receptor T (CAR T) cells: another cancer therapy with potential applications in kidney disease and transplantation? [J]. Kidney Int, 2018, 94(1): 4-6.
- [12] ALBINGER N, HARTMANN J, ULLRICH E. Current status and perspective of CAR-T and CAR-NK cell therapy trials in Germany [J]. Gene Ther, 2021, 28(9): 513-27.
- [13] MACKENSEN A, MULLER F, MOUGIAKAKOS D, et al. Anti-CD19 CAR T cell therapy for refractory systemic lupus erythematosus [J]. Nature medicine, 2022, 28(10): 2124-32.
- [14] MULLER F, TAUBMANN J, BUCCI L, et al. CD19 CAR T-Cell Therapy in Autoimmune Disease A Case Series with Follow-up [J]. N Engl J Med, 2024, 390(8): 687-700.
- [15] LI Y R, LYU Z, CHEN Y, et al. Frontiers in CAR-T cell therapy for autoimmune diseases [J]. Trends Pharmacol Sci, 2024, 45(9): 839-57.
- [16] YANG C, SUN C, TAN B, et al. Allogeneic anti-CD19 CAR-T cells induce remission in refractory systemic lupus erythematosus [J]. Cell Res, 2025.
- [17] WANG X, WU X, TAN B, et al. Allogeneic CD19-targeted CAR-T therapy in patients with severe myositis and systemic sclerosis [J]. Cell, 2024, 187(18): 4890-904 e9.
- [18] WANG W, HE S, ZHANG W, et al. BCMA-CD19 compound CAR T cells for systemic lupus erythematosus: a phase 1 open-label clinical trial [J]. Annals of the rheumatic diseases, 2024, 83(10): 1304-14.

- [19] HOXHA E, REINHARD L, STAHL R A K. Membranous nephropathy: new pathogenic mechanisms and their clinical implications [J]. Nature reviews Nephrology, 2022, 18(7): 466-78.
- [20] KOLLNER S M S, SEIFERT L, ZAHNER G, et al. Strategies Towards Antigen-Specific Treatments for Membranous Nephropathy [J]. Frontiers in immunology, 2022, 13: 822508.
- [21] LEE D W, SANTOMASSO B D, LOCKE F L, et al. ASTCT Consensus Grading for Cytokine Release Syndrome and Neurologic Toxicity Associated with Immune Effector Cells [J]. Biology of blood and marrow transplantation: journal of the American Society for Blood and Marrow Transplantation, 2019, 25(4): 625-38.
- [22] LEUKEMIA, LYMPHOMA GROUP C S O H C M A, GROUP OF HEMATOPOIETIC STEM CELL T, et al. [Consensus of Chinese experts on the clinical management of chimeric antigen receptor T-cell-associated neurotoxicity (2022)] [J]. Zhonghua Xue Ye Xue Za Zhi, 2022, 43(2): 96-101.